CLINICAL TRIAL: NCT05311683
Title: Work-related Musculoskeletal Disorder Between Egyptian Pediatric Dentists and General Dentists: A Cross Sectional Study
Brief Title: Work Related MSDs Between Egyptian Dentists
Acronym: MSDs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Mahmoud Madboly, Principle investigator, Cairo University
Other Study IDs: work related MSDs
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Musculoskeletal Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the musculoskeletal pain and discomfort among specialized pediatric dentists and general dentists.

DETAILED DESCRIPTION:
Musculoskeletal disorders are caused by the accumulation of mechanical and various stresses on the body, such as repetitive work of specific body parts, uncomfortable and unnatural work postures, high work intensity, excessive force, insufficient rest, cold working environment, and frequency. It is defined as musculoskeletal complaints, musculoskeletal pain that reflect a number of conditions, such as neck pain, back pain, shoulder pain, pain of limbs, carpal tunnel syndrome, myofacial dysfunction syndrome, atypical facial pain Although these musculoskeletal disorders can appear in all occupational groups, it is known that the incidence of musculoskeletal pain symptoms is higher in the dentist occupational group than in other occupational groups This is because dentists have to sit or stand for a long time and keep their head, neck, and shoulders in a fixed position for a long time.Bending motions, twisting motions, forward bent sitting postures, and relatively static working postures, which dentists mainly take during their treatment, are considered risk factors. According to a study on musculoskeletal disorders in Sharkia - low-back pain was the most prevalent musculoskeletal complaint that reported by (56.9%) of the subjects, followed by 50.4%, 47.2% and 42.3% complained of pain in the order of wrist, neck and shoulders Valachi and Valachi (2003) reported that approximately 81% of US dentists suffered from neck, shoulder and back pain Moreover, with the onset of the Covid-19 pandemic, the use of additional protective devices increases the mental stress, the risks of imbalanced postures and further reduces the freedom of movement.

Although there are many studies on musculoskeletal disorders in the dental profession, studies on pediatric dentistry are rare. In the case of pediatric dentists, the cooperation of young patients is insufficient, the treatment time is short, and they are exposed to various environments such as general anaesthesia . In addition, pediatric dental chairs do not fit children of all ages, which affects the attitude of dentists

ELIGIBILITY:
Inclusion Criteria:

* Graduated Egyptian dentists since 2015 , practicing in egypt since 2016
* Dentists Working hours more than 4 hours and at least 4 days per week
* Pediatric dentists treating one child at least per working day

Exclusion Criteria:

* Participants with history of serious trauma or fracture
* The presence of serious medical conditions or a transmissible disease such as malignant disease, hepatitis, AIDS etc.
* Participants will not sign the consent or complete the questionnaire.

Ages: 29 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study will be conducted in Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Egypt. The questionnaire will be provided to participants
  1. Through e-mail and an internet form to complete
  2. Handled personally to complete
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of (WMSDs) among Pediatric and General dentists | 1 year
  Numerical value

SECONDARY OUTCOMES:
Association between WMSDs and ergonomic assessment of their exposure to risk factor | 1 years
  Numerical value

CONTACTS AND LOCATIONS:
Overall Officials: Hala m Abbas, Professor, Study Director — Cairo U
Locations (1):
- Cairo university, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Karahan A, Kav S, Abbasoglu A, Dogan N. Low back pain: prevalence and associated risk factors among hospital staff. J Adv Nurs. 2009 Mar;65(3):516-24. doi: 10.1111/j.1365-2648.2008.04905.x. PMID 19222649
- [Background] Hales TR, Bernard BP. Epidemiology of work-related musculoskeletal disorders. Orthop Clin North Am. 1996 Oct;27(4):679-709. PMID 8823390
- [Background] Marshall ED, Duncombe LM, Robinson RQ, Kilbreath SL. Musculoskeletal symptoms in New South Wales dentists. Aust Dent J. 1997 Aug;42(4):240-6. doi: 10.1111/j.1834-7819.1997.tb00128.x. PMID 9316311
- [Background] Valachi B, Valachi K. Mechanisms leading to musculoskeletal disorders in dentistry. J Am Dent Assoc. 2003 Oct;134(10):1344-50. doi: 10.14219/jada.archive.2003.0048. PMID 14620013
- [Background] Barjatya K, Vatsal A, Kambalimath HV, Kulkarni VK, Reddy NB. Pediatric dental chair vs. traditional dental chair: a pediatric dentist's poll. J Indian Soc Pedod Prev Dent. 2015 Jan-Mar;33(1):35-9. doi: 10.4103/0970-4388.148973. PMID 25572371